CLINICAL TRIAL: NCT05688800
Title: Pressure Release Versus Thoracic Spine Manipulation in Rhomboids Myofascial Pain Syndrome
Brief Title: Pressure Release Versus Thoracic Manipulation in Rhomboids MPS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marwa Medhat Fawzy Mohamed, principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: p.t.REC/012/004127
Record Dates: First submitted 2023-01-09; First posted 2023-01-18 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Myofascial Pain Syndrome; Trigger Point Pain, Myofascial
Keywords: Myofascial pain syndrome; pressure release; Thoracic manipulation; Active trigger point; Rhomboids trigger point
MeSH Terms: conditions — Myofascial Pain Syndromes

STUDY DESIGN:
Intervention Model Description: Control group: will receive conventional physical therapy treatment Experimental group 1: will receive conventional physical therapy treatment in addition to pressure release Experimental group 2: will receive conventional physical therapy treatment in addition to thoracic spine manipulation
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Active Comparator): Each participant include 22 participants will receive conventional physical therapy treatment including TENS, continuous ultrasound ,infra-red radiation and combined stretching and strengthening exercise
  Interventions: Device: conventional therapy
- Experimental group 1 :pressure release technique (Experimental): Each participant include 22 participants will receive the conventional physical therapy treatment in addition to pressure release technique
  Interventions: Other: Experimental group 1 : pressure release technique
- Experimental group 2: thoracic spine manipulation (Experimental): Each participant include 22 participants will receive the conventional physical therapy treatment in addition to thoracic spine manipulation
  Interventions: Other: Experimental group 2: thoracic spine manipulation

INTERVENTIONS:
Device: conventional therapy — Participants in control group will receive conventional physical therapy treatment including Conventional TENS high frequency (90-130hz) low intensity according to the patient sensation for 30-45 min(Gozani, 2019) , continuous ultrasound with frequency 1 MHz and intensity 0.8 W/cm 2 will be applied by slow circular perpendicular movements with slightly deep pressure. Application time was 5 minutes at each side of the level of C7_T4 along the medial borders of the scapulae width, infra-red radiation will be four 15 minutes and directed perpendicular to the inter-scapular area, centered at the level of C7_T4 long and between the 2 medial borders of the scapulae width . Also combined stretching and strengthening exercise will be added due to its greater pain-relieving effect
  Arms: Control group
Other: Experimental group 1 : pressure release technique — Participants who are assigned to this group will receive conventionalphysical therapy treatment in addition to pressure release technique. the participant will be positioned either sitting or prone position according to his preferred position, the researcher will apply the pressure release procedure by a pressure below the PPT dependent onsoft tissue release. When the researcher detected a reduction in soft tissue resistance, the amount of compression will be increased. The pressure should -33- be nonpainful, applied at slow rate, and will maintained until release of tissue barrier. Further pressure was increased to reach a new barrier. The pressure will last 60 seconds. With the thumb or the second and third fingers, the non-painful manual therapy approach was applied to the active MTrPs of therhomboid muscle
  Arms: Experimental group 1 :pressure release technique
Other: Experimental group 2: thoracic spine manipulation — Thoracic spine manipulation will be performed as screw thrust manipulation technique; the vertebral transverse processes will beforced from posterior to anterior direction. The direction of the manipulation should be identified by applying springing test to the adjacent spinous process to determine the painful and stiff segment. Patient will be prone and researcher hand placement will be positioned as the following one pisiform on the right facet of the above, and the other pisiform on the left facet of the below vertebrae.A slack will be taken up. The thrust applied directly toward the patient once
  Arms: Experimental group 2: thoracic spine manipulation

SUMMARY:
The purpose of the stud will be to compare the effect of pressure release with thoracic spine manipulation on pain intensity level and pain pressure threshold, thoracic spine ROM and physical function onactive rhomboids muscle trigger point in myofascial pain syndrome.

DETAILED DESCRIPTION:
Myofascial pain syndrome (MPS) is one of the most common chronic disorders causing persistent musculoskeletal pain which is characterized by myofascial trigger points (MTrPs) in palpable taut bands of skeletal muscle. In recent years, due to our modern lifestyle people is exposed to postural stresses, inefficient biomechanics, repetitive postural dysfunction, which are some of the causes of myofascial pain syndrome .Active Rhomboid muscle trigger point are one of the main causes of inter- scapular pain, as the referral pattern of this muscle is on the medial border of the scapula. The aim of the study is to find if there any significant difference between the effect of pressure release and thoracic spine manipulation on pain intensity level, pain pressure threshold ,thoracic spine ROM and physical function and symptoms in people with musculoskeletal disorders of the upper limb on active rhomboids muscle trigger point in myofascial pain syndrome. 66 participants will be allocated randomly to three groups ; The Participants will be assigned randomly into three groups by simple methods of randomization. Control group: will receive conventional physical therapy treatment, Experimental group 1: will receive conventional physical therapy treatment in addition to pressure release Experimental group 2: will receive conventional physical therapy treatment in addition to thoracic spine manipulation.

ELIGIBILITY:
Inclusion Criteria:

Participants ages will be from 18 to 30 years Participants will be from both genders. Participants that have Myofascial pain syndrome due to at least one active trigger points in rhomboid muscle (Haleema and Riaz, 2021). Participants have myofascial pain syndrome since more than three months. Presence of a palpable taut band in a skeletal muscle

Exclusion Criteria:

Malignancy. Fractures of the Thoracic spine. Cervical radiculopathy or myelopathy. Vascular syndromes such as vertebrobasilar insufficiency. Rheumatoid arthritis. Neck or upper back surgery. Taking anticoagulants. Local infection. Whiplash injury. Open wounds. Pregnancy. Receiving radiation or chemotherapy. Scapular pain due to any degeneration disease. Osteoporosis. Cardiac pacemaker. Any contraindication for thoracic manipulation

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity level | up to three weeks
  pain intensity level will be measured by visual analogue scale (VAS)
Pressure Pain threshold level (PPT) | up to three weeks
  pressure pain threshold level (PPT) will be measured by digital algometer

SECONDARY OUTCOMES:
Rom of Motion | up to three weeks
  rom will be measured by digital inclinometer
Physical function | up to three weeks
  physical function will be measured by Disability of Arm, Shoulder, and Hand questionnaire (DASH)